CLINICAL TRIAL: NCT04824092
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial Comparing the Efficacy and Safety of Tafasitamab Plus Lenalidomide in Addition to R-CHOP Versus R-CHOP in Previously Untreated, High-intermediate and High-risk Patients With Newly-diagnosed Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Tafasitamab + Lenalidomide + R-CHOP Versus R-CHOP in Newly Diagnosed High-intermediate and High Risk DLBCL Patients
Acronym: frontMIND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOR208C310; 2022-500237-92-00 (Registry Identifier: EU CT Number); 2020-002990-84 (EudraCT Number)
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: DLBCL; CD19; monoclonal antibody; tafasitamab; lenalidomide; R-CHOP; Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tafasitamab; Lenalidomide; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tafasitamab plus lenalidomide in addition to R-CHOP (Experimental): Patients will receive tafasitamab plus lenalidomide in addition to R-CHOP for six 21-day cycles:
  Tafasitamab dose: 12 mg/kg body weight. Each 21-day cycle (cycles 1-6) will comprise of a tafasitamab IV infusion on Day 1, Day 8 and Day 15.
  Lenalidomide dose: 25 mg as a starting dose per os (orally) once per day on Days 1-10 of each 21-day cycle
  R-CHOP dose: Rituximab (or locally approved biosimilar) 375 mg/m2, IV Day 1 of every 21-day cycle; Cyclophosphamide 750 mg/m2, IV Day 1 of 21-day cycle; Doxorubicin 50 mg/m2, IV Day 1 of 21-day cycle; Vincristine 1.4 mg/m2 (max 2 mg) IV Day 1 of 21-day cycle; Prednisone/prednisolone 100 mg/day, per os, Day 1-5 of every 21-day cycle
  Interventions: Drug: Tafasitamab; Drug: Lenalidomide; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- Tafasitamab placebo plus lenalidomide placebo in addition to R-CHOP (Placebo Comparator): Patients will receive tafasitamab placebo plus lenalidomide placebo in addition to R-CHOP for six 21-day cycles:
  Tafasitamab placebo: 0.9% saline solution Days 1, 8 and 15 of each 21-day cycle
  Lenalidomide placebo: Days 1-10 of each 21-day cycle
  R-CHOP dose: Rituximab (or locally approved biosimilar) 375 mg/m2, IV Day 1 of every 21-day cycle; Cyclophosphamide 750 mg/m2, IV Day 1 of 21-day cycle; Doxorubicin 50 mg/m2, IV Day 1 of 21-day cycle; Vincristine 1.4 mg/m2 (max 2 mg) IV Day 1 of 21-day cycle; Prednisone/prednisolone 100 mg/day, per os, Day 1-5 of every 21-day cycle
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Tafasitamab placebo; Drug: Lenalidomide placebo

INTERVENTIONS:
Drug: Tafasitamab — Tafasitamab IV infusion will be administered as per the schedule specified in the respective arm.
  Other Names: Monjuvi
  Arms: Tafasitamab plus lenalidomide in addition to R-CHOP
Drug: Lenalidomide — Lenalidomide PO will be administered as per the schedule specified in the respective arm.
  Arms: Tafasitamab plus lenalidomide in addition to R-CHOP
Drug: Rituximab — Rituximab IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Cyclophosphamide — Cyclophosphamide IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Doxorubicin — Doxorubicin IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Vincristine — Vincristine IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Prednisone — Prednisone PO will be administered as per the schedule specified in the respective arm.
Drug: Tafasitamab placebo — 0.9% saline solution IV infusion will be administered as per the schedule specified in the respective arm.
  Arms: Tafasitamab placebo plus lenalidomide placebo in addition to R-CHOP
Drug: Lenalidomide placebo — Placebo matching to lenalidomide PO will be administered as per the schedule specified in the respective arm.
  Arms: Tafasitamab placebo plus lenalidomide placebo in addition to R-CHOP

SUMMARY:
This is a phase 3, multicenter, randomized, double-blind, placebo-controlled trial designed to compare the efficacy and safety of the humanized monoclonal anti CD19 antibody tafasitamab plus lenalidomide in addition to R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) versus R-CHOP in previously untreated, high-intermediate and high-risk patients with newly-diagnosed DLBCL

ELIGIBILITY:
Major Inclusion Criteria:

* Previously untreated patients with local biopsy-proven, CD20-positive DLBCL, including one of the following diagnoses by 2016 World Health Organization (WHO) classification of lymphoid neoplasms are eligible:

  1. DLBCL, NOS including GCB type, ABC type
  2. T-cell rich large BCL
  3. Epstein-Barr virus-positive DLBCL, NOS
  4. Anaplastic lymphoma kinase (ALK)-positive large BCL
  5. Human herpes virus-8 (HHV8)-positive DLBCL, NOS
  6. High-grade BCL with MYC and B-cell lymphoma 2 (BCL2) and/or B-cell lymphoma 6 (BCL6) rearrangements (double-hit or triple-hit lymphoma). Please note: Patients must be appropriate candidates for R-CHOP. If an investigator deems a patient with a known double- or triple-hit lymphoma (HGBL) should be treated more aggressively (e.g. dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab [DA-EPOCH-R] or cyclophosphamide, vincristine, doxorubicin and dexamethasone (CVAD) followed by methotrexate and cytarabine [Hyper CVAD]), this patient would not be considered eligible for this study
  7. HGBL-NOS
  8. DLBCL coexistent with either follicular lymphoma (FL) of any grade, gastric MALT lymphoma or non-gastric MALT lymphoma
  9. FL grade 3b
* Availability of archival or freshly collected tumor tissue sent for retrospective central pathology review
* IPI status of 3 to 5 (for patients > 60 years of age) or aaIPI 2 to 3 (for patients ≤ 60 years of age)
* Diagnosis to treatment interval, defined as the time between the date of DLBCL diagnosis (date of the first biopsy specimen containing B Cell lymphoma according to the local pathology report) and the start of treatment (C1D1) ≤ 28 days
* ECOG performance status of 0, 1, or 2
* Left ventricular ejection fraction equal to or greater 50% as assessed by local echocardiography or cardiac multi-gated acquisition (MUGA) scan
* Adequate hematologic function
* Female participants: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods and refrain from breast feeding and donating eggs; agreement to ongoing pregnancy testing during the course of the study, and after study therapy has ended
* Male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom and agreement to refrain from donating sperm

Major Exclusion Criteria:

* Any other histological type of lymphoma according to WHO 2016 classification of lymphoid neoplasms, e.g., primary mediastinal (thymic) large B-cell lymphoma, Burkitt's lymphoma, BCL, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma (grey-zone lymphoma); primary effusion lymphoma; primary cutaneous DLBCL, leg type; primary DLBCL of the CNS; DLBCL arising from CLL or indolent lymphoma
* History of prior non-hematologic malignancy except for the following:

  1. Malignancy treated with curative intent and with no evidence of active disease present for more than 2 years before screening
  2. Adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled non-melanomatous skin cancer
  3. Adequately treated carcinoma in situ without current evidence of disease
* Any systemic anti-lymphoma and/or investigational therapy prior to the start of C1D1, except for permitted pre-phase treatment
* Contraindication to any of the individual components of R-CHOP, including prior receipt of anthracyclines
* Known CNS lymphoma involvement
* Known active systemic bacterial, viral, fungal, or other infection at screening, including patients with suspected active or latent tuberculosis (as confirmed by a positive interferon-gamma release assay)
* History or evidence of clinically significant cardiovascular, CNS and/or other systemic disease that in the investigator's opinion would preclude participation in the study or compromise the patient's ability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 899 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS-INV | Time from date of randomization until Progressive Disease or death from any cause. In this trial, the primary endpoint is PFS as assessed by the investigator (up to 43 months)
  Progression-Free Survival as assessed by the investigator using the Lugano Response Criteria for Malignant Lymphoma

SECONDARY OUTCOMES:
EFS-INV | From randomization until the first occurrence of disease progression or relapse as assessed by the INV using, start of new anti-lymphoma treatment or death from any cause, whichever occurs first (up to 43 months)
  Event-Free Survival as assessed by the investigator using the Lugano Response Criteria for Malignant Lymphoma
OS | From randomization until the date of death from any cause (up to 62 months)
  Overall Survival
Metabolic PET-negative CR-rate at EOT by BIRC | End of treatment, 4-8 weeks after last dose
  Metabolic PET-negative CR rate defined as the proportion of patients who achieved metabolic PET-negative CR as per Lugano 2014 criteria based on PET/CTs performed at the end of the treatment by BIRC
Metabolic PET-negative CR-rate at EOT by INV | End of treatment, 4-8 weeks after last dose
  Metabolic PET-negative CR rate defined as the proportion of patients who achieved metabolic PET-negative CR as per Lugano 2014 criteria based on PET/CTs performed at the end of the treatment by the investigator
ORR as per INV at EOT | 6 ± 2 weeks after End of Treatment
  Overall response rate defined as the proportion of patients with CR or PR as per Lugano 2014 criteria based on assessment at the end of the treatment by the INV
Time to next anti-lymphoma treatment (TTNT) | From randomization date to start of next anti-lymphoma therapy (for any reason including disease progression, treatment toxicity, and patient preference) or death due to any cause, whatever comes first (up to 43 months)
  TTNT is defined as the time from randomization date to start of next anti-lymphoma therapy (for any reason including disease progression, treatment toxicity, and patient preference) or death due to any cause, whatever comes first.
Duration of Complete Response (CR) as assessed by the investigator | From the date of the first occurrence of a documented CR, to the date of progression, relapse, or death from any cause, whichever is earlier (up to 43 months)
  Duration of CR is defined as the time from the date of the first occurrence of a documented CR, to the date of progression, relapse, or death from any cause, whichever is earlier for the subgroup of patients with a Best Overall Response (BOR) of CR.
EFS at 3 years | 36 months after randomization
  Event-Free Survival as assessed by the investigator
PFS at 3 years | 36 months after randomization
  Progression-Free Survival as assessed by the investigator
OS at 3 years | 36 months after randomization
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Director, Study Director — Incyte Corporation
Locations (270):
- United States (47):
  - MorphoSys Research Site, Daphne, Alabama
  - MorphoSys Research Site, Anaheim, California
  - MorphoSys Research Site, Clovis, California
  - MorphoSys Research Site, Fullerton, California
  - MorphoSys Research Site, Harbor City, California
  - MorphoSys Research Site, Los Angeles, California
  - MorphoSys Research Site, San Diego, California
  - MorphoSys Research Site, Whittier, California
  - MorphoSys Research Site, Aurora, Colorado
  - MorphoSys Research Site, Jacksonville, Florida
  - MorphoSys Research Site, Honolulu, Hawaii
  - MorphoSys Research Site, Wichita, Kansas
  - MorphoSys Research Site, Lexington, Kentucky
  - MorphoSys Research Site, Louisville, Kentucky
  - MorphoSys Research Site, Baltimore, Maryland
  - MorphoSys Research Site, Bethesda, Maryland
  - MorphoSys Research Site, Columbia, Maryland
  - MorphoSys Research Site, Detroit, Michigan
  - MorphoSys Research Site, Minneapolis, Minnesota
  - MorphoSys Research Site, Rochester, Minnesota
  - MorphoSys Research Site, Kansas City, Missouri
  - MorphoSys Research Site, Lebanon, New Hampshire
  - MorphoSys Research Site, Florham Park, New Jersey
  - MorphoSys Research Site, Buffalo, New York
  - MorphoSys Research Site, Rochester, New York
  - MorphoSys Research Site, Canton, Ohio
  - MorphoSys Research Site, Cincinnati, Ohio
  - MorphoSys Research Site, Eugene, Oregon
  - MorphoSys Research Site, Danville, Pennsylvania
  - MorphoSys Research Site, Chattanooga, Tennessee
  - MorphoSys Research Site, Germantown, Tennessee
  - MorphoSys Research Site, Nashville, Tennessee
  - MorphoSys Research Site, Austin, Texas
  - MorphoSys Research Site, Bedford, Texas
  - MorphoSys Research Site, Denison, Texas
  - MorphoSys Research Site, Fort Worth, Texas
  - MorphoSys Research Site, Houston, Texas
  - MorphoSys Research Site, McAllen, Texas
  - MorphoSys Research Site, Tyler, Texas
  - MorphoSys Research Site, Ogden, Utah
  - MorphoSys Research Site, Salt Lake City, Utah
  - MorphoSys Research Site, Gainesville, Virginia
  - MorphoSys Research Site, Roanoke, Virginia
  - MorphoSys Research Site, Virginia Beach, Virginia
  - MorphoSys Research Site, Olympia, Washington
  - MorphoSys Research Site, Tacoma, Washington
  - MorphoSys Research Site, Marshfield, Wisconsin
- Argentina (4):
  - MorphoSys Research Site, Buenos Aires
  - MorphoSys Research Site, Cipolletti
  - MorphoSys Research Site, Rosario
  - MorphoSys Research Site, San Miguel de Tucumán
- Australia (26):
  - MorphoSys Research Site, Adelaide
  - MorphoSys Research Site, Ballarat
  - MorphoSys Research Site, Birtinya
  - MorphoSys Research Site, Brisbane
  - MorphoSys Research Site, Canberra
  - MorphoSys Research Site, Clayton
  - MorphoSys Research Site, Frankston
  - MorphoSys Research Site, Geelong
  - MorphoSys Research Site, Gold Coast
  - MorphoSys Research Site, Gosford
  - MorphoSys Research Site, Greenslopes
  - MorphoSys Research Site, Hobart
  - MorphoSys Research Site, Kingswood
  - MorphoSys Research Site, Kogarah
  - MorphoSys Research Site, Launceston
  - MorphoSys Research Site, Malvern
  - MorphoSys Research Site, Melbourne
  - MorphoSys Research Site, Nedlands
  - MorphoSys Research Site, Perth
  - MorphoSys Research Site, Richmond
  - MorphoSys Research Site, St Albans
  - MorphoSys Research Site, Sydney
  - MorphoSys Research Site, Townsville
  - MorphoSys Research Site, Wahroonga
  - MorphoSys Research Site, Waratah
  - MorphoSys Research Site, Wollongong
- Austria (5):
  - MorphoSys Research Site, Innsbruck
  - MorphoSys Research Site, Linz
  - MorphoSys Research Site, Rankweil
  - MorphoSys Research Site, Sankt Pölten
  - MorphoSys Research Site, Vienna
- Canada (5):
  - MorphoSys Research Site, Halifax
  - MorphoSys Research Site, London
  - MorphoSys Research Site, Montreal
  - MorphoSys Research Site, Saskatoon
  - MorphoSys Research Site, Sherbrooke
- Colombia (2):
  - MorphoSys Research Site, Medellín
  - MorphoSys Research Site, Valledupar
- Czechia (5):
  - MorphoSys Research Site, Brno
  - MorphoSys Research Site, Hradec Králové
  - MorphoSys Research Site, Olomouc
  - MorphoSys Research Site, Ostrava
  - MorphoSys Research Site, Prague
- France (16):
  - Morphosys Research Site, Caen, Cedex 9
  - Morphosys Research Site, Bordeau, Pessac Cedax
  - MorphoSys Research Site, Amiens
  - MorphoSys Research Site, Bordeaux
  - MorphoSys Research Site, La Tronche
  - Morphosys Research Site, Le Chesnay
  - MorphoSys Research Site, Le Mans
  - MorphoSys Research Site, Lille
  - MorphoSys Research Site, Limoges
  - MorphoSys Research Site, Marseille
  - MorphoSys Research Site, Nantes
  - MorphoSys Research Site, Poitiers
  - MorphoSys Research Site, Quimper
  - MorphoSys Research Site, Saint-Priest-en-Jarez
  - MorphoSys Research Site, Vandœuvre-lès-Nancy
  - MorphoSys Research Site, Vannes
- Germany (23):
  - MorphoSys Research Site, Aachen
  - MorphoSys Research Site, Augsburg
  - MorphoSys Research Site, Berlin
  - Morphosys Research Site, Berlin
  - MorphoSys Research Site, Bonn
  - MorphoSys Research Site, Chemnitz
  - MorphoSys Research Site, Cottbus
  - MorphoSys Research Site, Göttingen
  - MorphoSys Research Site, Halle
  - MorphoSys Research Site, Heilbronn
  - MorphoSys Research Site, Jena
  - MorphoSys Research Site, Kassel
  - MorphoSys Research Site, Lübeck
  - MorphoSys Research Site, Magdeburg
  - MorphoSys Research Site, Mainz
  - MorphoSys Research Site, Marburg
  - MorphoSys Research Site, Munich
  - MorphoSys Research Site, Münster
  - MorphoSys Research Site, Paderborn
  - MorphoSys Research Site, Tübingen
  - MorphoSys Research Site, Wiesbaden
  - MorphoSys Research Site, Wuppertal
  - MorphoSys Research Site, Würzburg
- Hungary (5):
  - MorphoSys Research Site, Budapest
  - MorphoSys Research Site, Debrecen
  - MorphoSys Research Site, Győr
  - Morphosys Research Site, Nyíregyháza
  - MorphoSys Research Site, Pécs
- Ireland (2):
  - MorphoSys Research Site, Dublin
  - MorphoSys Research Site, Limerick
- Israel (6):
  - MorphoSys Research Site, Beersheba
  - MorphoSys Research Site, Haifa
  - MorphoSys Research Site, Jerusalem
  - MorphoSys Research Site, Petah Tikva
  - Morphosys Research Site, Ramat Gan
  - MorphoSys Research Site, Tel Aviv
- Italy (21):
  - MorphoSys Research Site, Bergamo
  - MorphoSys Research Site, Brescia
  - MorphoSys Research Site, Candiolo
  - MorphoSys Research Site, Catania
  - MorphoSys Research Site, Forlì
  - MorphoSys Research Site, Genoa
  - MorphoSys Research Site, Lecce
  - MorphoSys Research Site, Milan
  - MorphoSys Research Site, Novara
  - MorphoSys Research Site, Orbassano
  - MorphoSys Research Site, Padua
  - MorphoSys Research Site, Palermo
  - MorphoSys Research Site, Pavia
  - MorphoSys Research Site, Ravenna
  - MorphoSys Research Site, Rimini
  - MorphoSys Research Site, Rozzano
  - MorphoSys Research Site, Siena
  - MorphoSys Research Site, Terni
  - MorphoSys Research Site, Tricase
  - MorphoSys Research Site, Trieste
  - MorphoSys Research Site, Turin
- Japan (14):
  - MorphoSys Research Site, Fukuoka
  - MorphoSys Research Site, Gifu
  - MorphoSys Research Site, Ibaraki
  - MorphoSys Research Site, Isehara
  - MorphoSys Research Site, Kagoshima
  - MorphoSys Research Site, Nagoya
  - MorphoSys Research Site, Narita-shi
  - MorphoSys Research Site, Okayama
  - MorphoSys Research Site, Osaka
  - MorphoSys Research Site, Osakasayama-shi
  - MorphoSys Research Site, Sapporo
  - MorphoSys Research Site, Tachikawa
  - MorphoSys Research Site, Tokyo
  - MorphoSys Research Site, Tsu
- Malaysia (11):
  - MorphoSys Research Site, Alor Star
  - MorphoSys Research Site, Ampang
  - MorphoSys Research Site, George Town
  - MorphoSys Research Site, Ipoh
  - MorphoSys Research Site, Johor Bahru
  - MorphoSys Research Site, Kota Bharu
  - MorphoSys Research Site, Kuala Lumpur
  - MorphoSys Research Site, Kuantan
  - MorphoSys Research Site, Kuching
  - MorphoSys Research Site, Petaling Jaya
  - MorphoSys Research Site, Subang Jaya
- MorphoSys Research Site, Auckland, New Zealand
- Philippines (3):
  - MorphoSys Research Site, Manila
  - MorphoSys Research Site, Pasig
  - MorphoSys Research Site, Quezon City
- Poland (2):
  - Morphosys Research Site, Lodz
  - MorphoSys Research Site, Warsaw
- Romania (6):
  - MorphoSys Research Site, Brasov
  - MorphoSys Research Site, Bucharest
  - Morphosys Research Site, Bucharest
  - Morphosys Research Site, Cluj-Napoca
  - Morphosys Research Site, Craiova
  - MorphoSys Research Site, Iași
- Russia (7):
  - MorphoSys Research Site, Kazan'
  - Morphosys Research Site, Moscow
  - MorphoSys Research Site, Novosibirsk
  - Morphosys Research Site, Petrozavodsk
  - MorphoSys Research Site, Saint Petersburg
  - Morphosys Research Site, Saint Petersburg
  - Morphosys research site, Ufa
- Serbia (3):
  - MorphoSys Research Site, Belgrade
  - MorphoSys Research Site, Kamenitz
  - Morphosys Research Site, Novi Sad
- Slovakia (2):
  - MorphoSys Research Site, Bratislava
  - MorphoSys Research Site, Košice
- South Korea (8):
  - MorphoSys Research Site, Busan
  - MorphoSys Research Site, Daegu
  - MorphoSys Research Site, Goyang-si
  - MorphoSys Research Site, Incheon
  - MorphoSys Research Site, Jeonju
  - MorphoSys Research Site, Jinju
  - MorphoSys Research Site, Seoul
  - MorphoSys Research Site, Yangsan
- Spain (11):
  - MorphoSys Research Site, Badalona
  - MorphoSys Research Site, Barcelona
  - MorphoSys Research Site, Girona
  - MorphoSys Research Site, Jerez de la Frontera
  - MorphoSys Research Site, Lugo
  - MorphoSys Research Site, Madrid
  - MorphoSys Research Site, Pamplona
  - MorphoSys Research Site, Salamanca
  - MorphoSys Research Site, Seville
  - MorphoSys Research Site, Valencia
  - MorphoSys Research Site, Vitoria-Gasteiz
- Taiwan (11):
  - Morphosys Research Site, Chang-hua
  - Morphosys Research Site, Chiayi City
  - Morphosys Research Site, Hualien City
  - MorphoSys Research Site, Kaohsiung City
  - Morphosys Research Site, Kaohsiung City
  - Morphosys Research Site, New Taipei City
  - Morphosys Research Site, Taichung
  - MorphoSys Research Site, Taichung
  - MorphoSys Research Site, Tainan
  - MorphoSys Research Site, Taipei
  - Morphsys Research Site, Taoyuan District
- Thailand (5):
  - MorphoSys Research Site, Bangkok
  - Morphosys Research Site, Bangkok
  - Morphosys Research Site, Chiang Mai
  - Morphosys Research Site, Khon Kaen
  - MorphoSys Research Site, Pathum Thani
- Turkey (Türkiye) (5):
  - MorphoSys Research Site, Ankara
  - MorphoSys Research Site, Izmir
  - MorphoSys Research Site, İzmit
  - MorphoSys Research Site, Malatya
  - MorphoSys Research Site, Mersin
- Ukraine (5):
  - Morphosys Research Site, Cherkasy
  - Morphosys Research Site, Chernihiv
  - Morphosys Research Site, Kharkiv
  - Morphosys Research Site, Kyiv
  - MorphoSys Research Site, Kyiv
- United Kingdom (9):
  - MorphoSys Research Site, Aberdeen
  - MorphoSys Research Site, Bath
  - MorphoSys Research Site, Birmingham
  - MorphoSys Research Site, Bristol
  - MorphoSys Research Site, London
  - Morphosys Research Site, London
  - MorphoSys Research Site, Nottingham
  - MorphoSys Research Site, Sutton
  - MorphoSys Research Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jelicic J, Juul-Jensen K, Bukumiric Z, Runason Simonsen M, Roost Clausen M, Ludvigsen Al-Mashhadi A, Schou Pedersen R, Poulsen CB, Gang AO, Brown P, El-Galaly TC, Stauffer Larsen T. International Prognostic Models as Tools for Selection of Higher-risk Trial-eligible Patients With Diffuse Large B-Cell lymphoma. Clin Lymphoma Myeloma Leuk. 2026 Jan;26(1):e62-e76. doi: 10.1016/j.clml.2025.08.020. Epub 2025 Sep 3. PMID 40993016
- [Derived] Belada D, Kopeckova K, Bergua Burgues JM, Stevens D, Andre M, Persona EP, Pichler P, Staber PB, Trneny M, Duell J, Waldron-Lynch M, Wagner S, Mukhopadhyay A, Dirnberger-Hertweck M, Burke JM, Nowakowski GS. Safety and efficacy of tafasitamab with or without lenalidomide added to first-line R-CHOP for DLBCL: the phase 1b First-MIND study. Blood. 2023 Oct 19;142(16):1348-1358. doi: 10.1182/blood.2023020637. PMID 37369099